CLINICAL TRIAL: NCT06164873
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study Evaluating the Efficacy and Safety of IBI362 9 mg in Chinese Participants With Obesity (GLORY-2)
Brief Title: A Study of IBI362 9 mg in Chinese Adults With Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI362B302
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- IBI362 (Experimental)
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: IBI362 — Once-weekly injections of gradually increased doses of IBI362
  Arms: IBI362
Drug: Placebo — Once-weekly injections of volume-matched placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase 3 clinical study evaluating the efficacy and safety of IBI362 9 mg in obese subjects. Subjects will be randomly assigned to IBI362 9 mg and placebo groups. All study treatment will be administered once-weekly and subcutaneously. The entire trial cycle includes a 2-week screening period, a 60-week double-blind treatment period, and a 12-week drug withdrawal follow-up period after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older at the time of signing informed consent
* Have a BMI ≥30 kg/m2
* Have a history of at least one self-reported unsuccessful dietary effort to lose body weight

For subjects with T2D at screening:

* Have a diagnosis of T2D according to the WHO classification above or equal to 3 months prior to the day of screening
* Treated with either diet and excercise alone or on stable treatment with up to 3 oral antidiabetic medications alone or in any combination (EXCEPT GLP-1R agonists or DPP-4 inhibitors) for at least 2 months prior to the day of screening
* HbA1c 7.0-10.0% (both inclusive) at screening
* Fasting blood glucose ≤11.1 mmol/L at screening

Exclusion Criteria:

• A self-reported change in body weight above 5% within 3 months before screening

For subjects without T2D at screening:

• HbA1c ≥6.5% as measured by local laboratory at screening

For subjects with T2D at screening:

* Have history of proliferative diabetic retinopathy, diabetic macular edema or non-proliferative diabetic retinopathy that required acute treatment
* Have had 2 or more episodes of ketoacidosis, hyperosmolar state or lactic acidosis within 6 months before screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Week 60
Proportion of Participants who Achieve ≥5% Body Weight Reduction | Week 60

SECONDARY OUTCOMES:
Proportion of Participants who Achieve ≥10% Body Weight Reduction | Week 60
Proportion of Participants who Achieve ≥15% Body Weight Reduction | Week 60
Proportion of Participants who Achieve ≥20% Body Weight Reduction | Week 60
Change from Baseline in Waist Circumference | Week 60
Change from Baseline in Systolic Blood Pressure | Week 60
Percent Change from Baseline in Triglycerides | Week 60
Percent Change from Baseline in non-high-density lipoprotein cholesteroal | Week 60
Percent Change from Baseline in low-density lipoprotein cholesterol | Week 60

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No